CLINICAL TRIAL: NCT06517680
Title: Efficacy of Tight Treatment in Rotator Cuff Tendinopathy Rotator Cuff Tendinopathy: a Randomized Controlled Trial Versus Standard Standard Management
Brief Title: Tight Control for Rotator Cuff Tendinopathy
Acronym: GREAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC23_0421
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: Rotator cuff tendinopathy, tight control, injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tight control group (Experimental): Patients will be seen every month for the first 3 months of follow-up During these consultations, shoulder pain and function will be assessed. Treatment adjustments (steroid injections, drugs and physiotherapy) will be proposed in line with predefined objectives.
  Interventions: Other: tight control management
- Control group (Active Comparator): Patients will have the usual follow-up for this indication, i.e. a follow-up consultation 3 months after the 1st consultation with the rheumatologist to assess their clinical course.
  Interventions: Other: standard follow-up

INTERVENTIONS:
Other: tight control management — Patients will be seen every month for the first 3 months of follow-up During these consultations, shoulder pain and function will be assessed. Treatment adjustments (steroid injections, drugs and physiotherapy) will be proposed in line with predefined objectives.
  Arms: Tight control group
Other: standard follow-up — Patients are monitored according to standard practice
  Arms: Control group

SUMMARY:
The main objective of the study is to determine whether tight management of patients in early rotator cuff tendinopathy would lead to better clinical improvement than standard management. In a randomized study, we propose to compare two types of management, with a tight control group having one consultation per month for the first 3 months, in order to readapt or intensify management, whereas the control group will only be seen at 3 months after inclusion. We hypothesize that this close follow-up will lead to more rapid clinical improvement and reduce the transition to chronicity and the associated costs (inclusion of a medico-economic analysis taking into account, in particular, healthcare consumption and time off work).

DETAILED DESCRIPTION:
Shoulder pain is a frequent reason for consultation, with a lifetime prevalence of 67%. Every year, around 1% of adults over 45 consult primary care because of shoulder pain. Of these, rotator cuff disorders account for around 70%. Pain associated with limited function has an impact on activities of daily living, and on professional activities, since the peak prevalence is between the ages of 45 and 64. They also represent a very costly problem, given the repeated absences from work they entail. Musculoskeletal disorders recognized as occupational illnesses are on the rise, with over 42,000 cases reported in France in 2012, 32% of them involving the shoulder. In 2006, the disease was estimated to have caused the loss of 7 million working days. A Swedish study also showed that the cost associated with painful shoulders was mainly represented by sick leave (84%).

Management of rotator cuff disorders initially involves symptomatic drug therapy (painkillers and non-steroidal anti-inflammatories), combined with rest and rehabilitation. Then, in case of insufficient improvement, subacromial steroid injection is often proposed. Despite the frequency of the condition, there are no established recommendations for the management of these patients. However, a recent study showed that the combination of posture advice and subacromial steroid injection was a more cost-effective strategy than either physiotherapy alone or infiltration alone. When we look at patients' outcome, chronic pain and impaired function are frequently seen, since 30-50% of patients still have symptoms after 1-2 years. It is therefore important to optimize the medical management of these patients, especially as at the stage of tendinopathy without rupture because surgical management is not always able to provide clinically significant benefits in terms of pain, function or quality of life.

In some chronic diseases, such as rheumatoid arthritis, it has been shown that early and tight control leads to better clinical results, as treatments are regularly and closely adapted to predefined objectives (remission or low disease activity). A significant improvement was also observed in diabetic patients under tight control leading to reduction in the risk of progression of retinal and neurological complications and significantly decreased risk of cardiovascular events.

The GREAT protocol is a prospective, randomized, multicenter study comparing two groups of patients:

* In the experimental or "tight control" group, patients will be seen every month for the first 3 months of follow-up. During these consultations, shoulder pain and function will be assessed. Treatment adjustments will be proposed in line with predefined objectives.
* In the control group, patients will have the usual follow-up for this indication, i.e. a follow-up consultation 3 months after the 1st consultation with the rheumatologist to assess their clinical course.

ELIGIBILITY:
Inclusion Criteria :

Patient with new-onset shoulder pain related to rotator cuff tendinopathy

* Age between 18 and 65
* Shoulder pain on activity for less than 6 months with VAS≥4/10 and/or OSS≥20
* Pain compatible with rotator cuff tendinopathy according to the rotator cuff tendinopathy according to the BESS (British Elbow and Shoulder Society) guidelines

Exclusion Criteria:

* Contraindication to steroid injections
* Shoulder pain related to trauma (dislocation, fracture) or acute tendon rupture requiring short-term surgery
* Steroid injection already performed on the shoulder studied for the current episode
* Neurological pathology affecting the shoulder
* Other shoulder disorders (inflammatory arthritis, frozen shoulder, glenohumeral joint instability, pain associated with acromioclavicular arthropathy)
* Tendon calcification > 0.5 cm.
* Previous shoulder surgery
* Full-thickness tear of one tendon
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-11-25 (Estimated); Study Completion 2027-11-25 (Estimated)

PRIMARY OUTCOMES:
Oxford Shoulder Score | 6 months
  Functional score including 12 items rated between 0 and 4 (total score/48) (best score = 48)

SECONDARY OUTCOMES:
Oxford Shoulder Score | 3 months and 12 months
  Functional score including 12 items rated between 0 and 4 (total score/48) (best score = 48)
pain at motion | 3 Months, 6 months, 12 months
  Visual Analogic Scale / 100 mm
Pain Self-Efficacy Questionnaire | 3 Months, 6 months, 12 months
  10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain.
Insomnia Severity Index | 3 Months, 6 months, 12 months
  7 item auto-questionnaire
number of shoulder surgeries | 12 months
  patients requiring shoulder surgery to manage their shoulder pain and/or disability
medico-economic study | 12 months
  Incremental cost-utility ratio (cost per QALY, Quality- Adjusted Life-Years)

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU Angers, Angers
  - CHU de Brest, Brest
  - CHRU de Tours, Chambray-lès-Tours
  - CH Cholet, Cholet
  - CH Vendée, La Roche-sur-Yon
  - CH du Mans, Le Mans
  - CHU de Nantes, Nantes
  - Chotard Emilie, Rennes

IPD SHARING:
Plan to Share IPD: Undecided